CLINICAL TRIAL: NCT01730092
Title: A Natural History Study of Novel Biomarkers in Pulmonary Arterial Hypertension
Brief Title: Natural History Study of Biomarkers in Pulmonary Arterial Hypertension
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130012; 13-CC-0012
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-19

CONDITIONS: Pulmonary Disease; Pulmonary Hypertension
Keywords: Vascular Inflammation; Microarray; Right Ventricular Function; Endothelial Dysfunction; Magnetic Resonance Imaging; Natural History
MeSH Terms: conditions — Lung Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Enroll up to 120 healthy volunteers, in order to obtain approximately 55 evaluable healthy volunteers matched to pulmonary arterial hypertension subjects for age and sex
- Pulmonary Arterial Hypertension Subjects: 150 subjects with pulmonary arterial hypertension; male or female, age grater than or equal to 18 99 years

SUMMARY:
Background:

- High blood pressure in the lungs, known as pulmonary arterial hypertension (PAH), is a rare disorder. Some people have disease-associated PAH and some have PAH from an unknown cause. Researchers want to follow the natural history of all PAH patients to understand how PAH progresses in order to discover targets for future research into new treatments. To further identify treatment targets, they will compare healthy volunteers to patients with PAH.

Objectives:

- To study the natural history of PAH.

Eligibility:

* Individuals at least 18 years of age who have PAH.
* Healthy volunteers at least 18 years of age.

Design:

* Participants with PAH will have periodic visits to the National Institutes of Health Clinical Center. After the first visit, they will return in 6 months and then yearly or every other year for as long as the study continues.
* The first visit will take up to 3 days. It will involve the following tests:
* Physical exam and medical history
* Blood and urine samples
* Heart and lung function tests and imaging studies
* Six-minute walk test
* Questions about exercise and physical activity
* Healthy volunteers will have only one visit to the Clinical Center, during which they will undergo screening tests, and complete many of the same tests as patients with PAH

DETAILED DESCRIPTION:
Introduction:

Pulmonary arterial hypertension (PAH) is a rare disorder associated with poor survival. Endothelial dysfunction resulting from 1) genetic susceptibility, and 2) a triggering stimulus that initiates pulmonary vascular injury, the two-hit hypothesis, appears to play a central role both in the pathogenesis and progression of PAH. Inflammation appears to drive this dysfunctional endothelial phenotype, propagating cycles of injury and repair in genetically susceptible patients with idiopathic PAH (IPAH) and patients with disease-associated PAH. However, despite mounting evidence of vascular inflammation in patients with PAH, detailed phenotypic studies are lacking on the temporal evolution of this process and its contribution to right ventricular (RV) and pulmonary vascular remodeling. We hypothesize that a detailed characterization of the temporal evolution of vascular inflammation in PAH and its impact on RV and pulmonary vascular function will add prognostic value to traditional measures of disease severity and suggest novel therapeutic targets for future research.

Objectives:

Patients with IPAH and disease-associated PAH will be recruited to the NIH and enrolled in this natural history study investigating the ability of circulating markers of vascular inflammation as well as high-resolution cardiac magnetic resonance imaging (MRI) to accurately stage severity of disease and/or predict clinically relevant outcomes.

Methods:

The total population for the study will be 150 PAH subjects and approximately 55 age and sex matched controls (i.e. each healthy volunteer is matched to less than or equal to 3 PAH subjects).

PAH subjects will undergo 1) standard clinical examinations including 6-minute walk distance and echocardiography; 2) cardiopulmonary exercise testing; 3) markers of coagulation and fibrotic disease; 4) plasma profiling of inflammatory

markers; 5) gene expression profiling of peripheral blood mononuclear cells PBMCs); 6) high-resolution MRI-based determination of pulmonary vascularand RV structure and function and 7) Cardiac CT scan.

Plasma markers of endothelial inflammation, PBMC expression profiles, and high-resolution cardiac MRI will also be studied in age and sex matched controls to define normal ranges and variability for each of these novel assessments. Comparison of these results to PAH subjects at baseline will be used to determine the degree to which these investigative tests distinguish PAH patients from healthy subjects. Likewise, baseline clinical evaluations of PAH subjects will be used to examine whether any novel test (inflammatory markers, or cardiac MRI), accurately classifies patients according to their disease severity. In addition, these tests will be investigated prospectively for their ability to predict PAH disease progression. Disease progression will be defined prospectively as a decrease in the 6-minute walk distance of greater than or equal to10 percent from baseline or clinical worsening requiring an escalation in therapy, hospitalization due to right heart failure, transplantation or death.

Additional plasma will be collected from PAH subjects and age/sex matched control subjects. This material will be used to probe for new biomarkers and inflammatory factors using discovery based approaches (i.e. Proteomics and pulmonary artery endothelial cell bioassay).

ELIGIBILITY:
* ELIGIBILITY:

The study will enroll subjects with confirmed and suspected NYHA/WHO Group 1 PH (68) as well as age and sex matched control subjects. Subjects must be at least 18 years of age and must be able to provide informed, written consent for participation in this study. There is no exclusion based on race or sex.

INCLUSION AND EXCLUSION CRITERIA FOR PAH SUBJECTS:

Inclusion Criteria:

The following parameters on RHC are required to meet the hemodynamic definition of PAH (NYHA/WHO Group I PH):

* mean pulmonary artery pressure of greater than 25 mmHg at rest,
* pulmonary capillary wedge pressure of less than or equal to 15 mmHg (or a left ventricular end-diastolic pressure of less than or equal to 12mmHg) and
* pulmonary vascular resistance of greater than 3 Wood units (240 dyn s cm(-5)).

For patients with suspected PAH (Group I PH) who have not undergone a RHC and/or additional testing to confirm the diagnosis, this testing will be completed as clinically indicated under a procedural consent. If clinically indicated (diagnostic) testing indicates that the subject with suspected PAH does not in fact meet standard criteria for PAH (Group I PH), then the subject will be removed from the study.

Exclusion Criteria:

* Pregnant or breastfeeding women (all women of childbearing potential will be required to have a screening urine or blood pregnancy test)
* Age less than 18 years
* Inability to provide informed written consent for participation in the study

INCLUSION AND EXCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS:

Inclusion Criteria for Control Subjects

Any healthy man or woman who is the appropriate age and sex for matching to a PAH patient

* Must be eligible for MRI and Gadolinium Based MRI studies
* Must be eligible for CT and Iodine Based Contrast CT studies

Exclusion Criteria for Healthy Control Subjects

* Current pregnancy or breastfeeding (All women of childbearing potential will be required to have a screening urine or blood pregnancy test)
* Electrocardiographic evidence of clinically relevant heart disease
* Symptoms of coronary or cardiac insufficiency
* More than one major risk factor for coronary artery disease (excluding age and sex)
* Obesity (defined as a body mass index > 30 kg/m^2)
* History of underlying conditions/risk factors associated with pulmonary hypertension such as collagen vascular disease, HIV infection, use of appetite suppressants, chronic liver disease or cirrhosis of the liver, chronic thromboembolic disease, congenital heart defects, hypoxemia and/or significant pulmonary parenchymal disease
* Systemic hypertension that is not well controlled (i.e. blood pressure at the time of screening greater than or equal to140/90 mmHg) in adults < 60 years old or greater than or equal to 150/90 mmHg in adults 60 years or older) on medications. Subjects taking > 2 anti-hypertensive medications will be excluded irrespective of their current blood pressure at time of screening
* Anemia, thrombocytopenia or coagulopathy
* Renal insufficiency (defined as an estimated glomerular filtration rate of < 60 mL/min/1.73m^2 of body surface area)
* Active tobacco use (> 6 months) in the past ten years, any tobacco use within 3 months prior to the screening evaluation or any tobacco use prior to completion of the study
* Inability to provide informed written consent for participation in the study
* History of recreational drug use with the exception of marijuana (as long as marijuana use was > 3 months from the time of study screening).

  * Volunteers may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer.

Exclusion Criteria for MRI in Healthy Control Subjects and Subjects with PAH

These contraindications include but are not limited to the following devices or conditions:

1. Implanted cardiac pacemaker or defibrillator
2. Cochlear Implants
3. Ocular foreign body (e.g. metal shavings)
4. Embedded shrapnel fragments
5. Central nervous system aneurysm clips
6. Implanted neural stimulator
7. Any implanted device that is incompatible with MRI
8. Unsatisfactory performance status as judged by the referring physician such that the subject could not tolerate an MRI scan. Examples of medical conditions that would not be accepted would include unstable angina and severe dyspnea at rest
9. Subjects requiring monitored sedation for MRI studies
10. Subjects with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.)
11. Subjects with severe back-pain or motion disorders who will be unable to tolerate supine positioning within the MRI scanner and hold still for the duration of the examination.

Exclusion Criteria for Gadolinium Based MRI Studies Only:

1. History of severe allergic reaction to gadolinium contrast agents despite pre- medication with diphenhydramine and prednisone
2. Chronic kidney disease (an estimated glomerular filtration rate of < 60 mL/min/1.73m^2 of body surface area)

Exclusion Criteria for Cardiac Computed Tomography in Healthy Control Subjects and Subjects with PAH:

1) Subjects with a condition precluding entry into the scanner (e.g. morbid

obesity, claustrophobia, etc.)

Exclusion Criteria for Iodine Based Contrast CTA Studies Only:

1. Serum creatinine > 1.4 mg/dL
2. History of multiple myeloma
3. Use of metformin-containing products less than 24 hours prior to contrast administration
4. History of significant allergic reaction to CTA contrast agents despite premedication with diphenhydramine and prednisone

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary clinical for PAH and community sample for controls
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2013-07-15 (Actual); Primary Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine whether any novel test (inflammatory markers or high resolution cardiac MRI), accurately classifies PAH subjects according to disease severity as assessed by their baseline 6-minute walk distance. | 10 years
  Compare outcomes in PAH subjects with controls

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Solomon, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Badesch DB, Raskob GE, Elliott CG, Krichman AM, Farber HW, Frost AE, Barst RJ, Benza RL, Liou TG, Turner M, Giles S, Feldkircher K, Miller DP, McGoon MD. Pulmonary arterial hypertension: baseline characteristics from the REVEAL Registry. Chest. 2010 Feb;137(2):376-87. doi: 10.1378/chest.09-1140. Epub 2009 Oct 16. PMID 19837821
- [Background] Rubin LJ. Primary pulmonary hypertension. Chest. 1993 Jul;104(1):236-50. doi: 10.1378/chest.104.1.236. No abstract available. PMID 8325077
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-CC-0012.html